CLINICAL TRIAL: NCT06401122
Title: Comparison of Dyslipidemia Among Diabetics Versus Non Diabetics in Haemodialysis
Brief Title: Comparison of Dyslipidemia Among Diabetics Versus Non Diabetics in Haemodialysis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Ali Abudeif Zaharn, doctor, Assiut University
Other Study IDs: Dyslipidemia haemodialysis
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Dyslipidemias
Keywords: haemodialysis diabetes mellitus
MeSH Terms: conditions — Dyslipidemias | interventions — Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic dialysis patients: fifty diabetic patients on regular haemodialysis more than 6 months
  Interventions: Procedure: haemodialysis
- Non-diabetic dialysis patients: fifty Non-diabetic patients on regular haemodialysis more than 6 months
  Interventions: Procedure: haemodialysis

INTERVENTIONS:
Procedure: haemodialysis — process of filtering the blood of a person whose kidneys are not working normally from uremic toxins

SUMMARY:
* How dyslipidemia common among Diabetic and non- Diabetic Haemodialysis patients.
* How differ dyslipidemia types among Diabetic and non- Diabetic in Haemodialysis patients. (Qualitative difference).

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a metabolic disease , a consequence of defects in insulin action, secretion, or both, and there are complications associated with it, such as nephropathy, retinopathy, neuropathy, cardiovascular complications ,cerebrovascular and peripheral arterial disease. Diabetic nephropathy, which occurs in about one third of type 2 diabetic patients, is the most common factor leading to end-stage renal disease (ESRD) . A very common metabolic abnormality associated with diabetes is dyslipidemia, which is characterized by a spectrum of quantitative and qualitative changes in lipids and lipoproteinsSeveral previous studies have pursued linking blood glucose levels to serum lipid activities. The etiology of dyslipidemia appears to be centered on the increased large TAG-rich very low-density lipoprotein-cholesterol (VLDL-C) and its impaired clearance. American diabetic association (ADA) defines dyslipidemia as hypercholesterolemia ≥200 mg/dl of serum total cholesterol, hypertriglyceridemia ≥150 mg/dl of serum triglyceride, reduced high density lipoprotein cholesterol (HDL-C) <40 mg/dl for men and <50 mg/dl for women, elevated low density lipoprotein cholesterol (LDL-C) ≥70 mg/dl and high TC to HDL-C ratio of ≥4.5. Normal plasma lipids and lipoprotein metabolism is critical for cellular cholesterol homeostasis and protection against atherosclerosis, renal disease and other complication . A study found that people with high blood pressure and overweight or obesity have a higher risk of developing dyslipidemia ,Early detection and effective control of blood lipid levels can reduce the morbidity and mortality of CVD in patients with DM. Therefore, it is important to determine the factors associated with dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 60 years.
* Patients undergoing regular conventional Haemodialysis for more than 6 months

Exclusion Criteria:

* Peritoneal Dialysis
* Haemodiafilteration
* Acute Kidney Injury
* Nephrotic syndrome
* Hypothyroidism
* Familial hypertriglyceridemia.
* Acute pancreatitis
* Connective tissue disease.
* Decompensated liver disease
* Active malignancy.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: haemodialysis patients for more than six months, and is with diabetes related to affect prevalance of dyslipidemia among these patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
dyslipidemia prevalence among Diabetic versus non- Diabetic Haemodialysis patients | baseline
  haemodialysis patients for more than six months, and is with diabetes related to affect prevalance of dyslipidemia among these patients

CONTACTS AND LOCATIONS:
Overall Officials: Salwa S. Elgendi, professor, Study Director — Assiut University; Essam M. Abdel-Aziz, doctor, Study Director — Assiut University

REFERENCES:
- [Background] Biadgo B, Abebe SM, Baynes HW, Yesuf M, Alemu A, Abebe M. Correlation between Serum Lipid Profile with Anthropometric and Clinical Variables in Patients with Type 2 Diabetes Mellitus. Ethiop J Health Sci. 2017 May;27(3):215-226. doi: 10.4314/ejhs.v27i3.3. PMID 29217920
- [Background] Zheng Y, Ley SH, Hu FB. Global aetiology and epidemiology of type 2 diabetes mellitus and its complications. Nat Rev Endocrinol. 2018 Feb;14(2):88-98. doi: 10.1038/nrendo.2017.151. Epub 2017 Dec 8. PMID 29219149
- [Background] Ariyanti R, Besral B. Dyslipidemia Associated with Hypertension Increases the Risks for Coronary Heart Disease: A Case-Control Study in Harapan Kita Hospital, National Cardiovascular Center, Jakarta. J Lipids. 2019 Apr 30;2019:2517013. doi: 10.1155/2019/2517013. eCollection 2019. PMID 31183219
- [Background] Hasan YK, Alsultan M, Anan MT, Hassn Q, Basha K. The prevalence of dyslipidemia in patients on hemodialysis: a cross-sectional study from Syria. Ann Med Surg (Lond). 2023 Jun 5;85(8):3838-3844. doi: 10.1097/MS9.0000000000000931. eCollection 2023 Aug. PMID 37554881